CLINICAL TRIAL: NCT06588153
Title: A Phase 4 Single-arm Open-label Study for the Efficacy and Safety of Prolia® in Participants With Glucocorticoid-induced Osteoporosis in Mainland China
Brief Title: A Study for the Evaluation of Efficacy and Safety of Prolia® in Participants With Glucocorticoid-induced Osteoporosis in Mainland China
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210125
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glucocorticoid-induced Osteoporosis
Keywords: Prolia®; Denosumab
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolia® (Experimental): Participants with glucocorticoid-induced osteoporosis (GIOP) will receive Prolia® every 6 months (Q6M).
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: Prolia® — Subcutaneous (SC) injection in pre-filled syringe.
  Other Names: Denosumab

SUMMARY:
The main objective of this study is to evaluate the efficacy of Prolia® in improving bone mass density (BMD) of lumbar spine at month 12.

ELIGIBILITY:
Inclusion Criteria

* Participant has provided informed consent prior to initiation of any study-specific activities/procedures.
* Male and female participants aged ≥ 18 years at the time of signing the informed consent.
* Participants are receiving glucocorticoid treatment at screening.
* Participants who are ≥ 50 years of age at the time of screening will be required to have a T-score with:

  - a BMD value equivalent to a T-score ≤ -2.5 at the lumbar spine or total hip or femoral neck; OR

  - a BMD value equivalent to a T-score ≤ -1.0 at the lumbar spine or total hip or femoral neck AND a history of osteoporotic fracture.
* Participants who are < 50 years of age at the time of screening will be required to have a T-score with a BMD value equivalent to a T-score ≤ -1.0 at the lumbar spine or total hip or femoral neck AND have a history of osteoporotic fracture.
* At least 2 lumbar vertebrae from L1 through L4 and 1 hip must be evaluable by dual-energy x-ray absorptiometry (DXA).
* Adequate organ function, defined as follows:

  * Hematological function:

    1. Absolute neutrophil count ≥ 1 x 10^9 /L
    2. Platelet count ≥ 100 x 10^9 /L
    3. Hemoglobin > 9 g/dL (90 g/L).
  * Coagulation function:

    1 Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time or activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN). Participants on chronic anticoagulation therapy who do not meet the criteria above may be eligible to enroll at the investigator's discretion per local standard of care.
  * Renal function:

    1 Estimated glomerular filtration rate based on Modification of Diet in Renal Disease (MDRD) calculation > 30 mL/min/1.73 m^2.
  * Hepatic function:

    1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase < 3 x ULN
    2. Total bilirubin (TBL) < 1.5 x ULN.

Exclusion Criteria

Disease Related

* Received other osteoporosis treatment or bone-active treatment with:

  - prior use of bisphosphonate:
  1. bisphosphonate use within 1 year unless duration of oral bisphosphonates treatment < 3 months use prior to screening
  2. administration of intravenous zoledronate within 2 years or intravenous bisphosphonate other than zoledronate within the last year.

     * fluoride or strontium for osteoporosis within the last 5 years
     * anabolic agents to include PTH or PTH derivatives within the last year
     * any prior use of products containing denosumab
* Administration of any of the following treatments within 3 months of screening:

  - any selective estrogen receptor modulator (estrogen agonist antagonist)
  * tibolone
  * anabolic steroids
  * testosterone above normal replacement doses not on stable dose
  * systemic hormone replacement therapy not on stable dose
  * systemic hormonal contraception not specified in the protocol or not on stable dose
  * calcitonin.
* Other bone-active drugs including:

  * anti-convulsants (except benzodiazepines) and heparin (low molecular weight heparin is allowed)
  * chronic systemic ketoconazole, androgens, adrenocorticotropic hormone (ACTH), cinacalcet, aluminum, lithium, protease inhibitors, gonadotropin-releasing hormone agonists.
* Any pretrial initiation of anti-inflammatory disease-modifying anti-rheumatic drug (DMARD) that is not consistent with the local Chinese label or guidelines.
* Participant has an active infection or history of infections as follows:

  * any active infection for which systemic anti-infectives were used within 4 weeks prior to screening
  * a serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to screening
  * recurrent or chronic infections or other active infection that, in the opinion of the investigator, might compromise the safety of the participant.

Other Medical Conditions

* History of hyperthyroidism (stable on antithyroid therapy is allowed) when suggested by medical history
* History of hypothyroidism (stable on thyroid replacement therapy is allowed) when suggested by medical history
* History of hypo- or hyperparathyroidism
* History of Addison's disease
* History of osteomalacia
* History of osteonecrosis of the jaw (ONJ)
* History of tooth extraction or other dental surgery within the prior 6 months
* Invasive dental work (per local oral surgeon's assessment) planned in the next 12 months
* History of Paget's disease of bone
* Other bone diseases which affect bone metabolism (e.g., osteopetrosis, osteogenesis imperfecta) (chart review)
* Received any solid organ or bone marrow transplant
* Known to have tested positive for human immunodeficiency virus, hepatitis C virus, hepatitis B surface antigen
* Participants with a history of any cancer (cured basal cell or squamous cell cancers are allowed)

Prior/Concurrent Clinical Study Experience • Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives, whichever is longer, since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Diagnostic Assessments

* Abnormalities of the following per central laboratory reference ranges:

  - Vitamin D deficiency (25[OH] vitamin D level < 20 ng/mL [< 49.9 nmol/L]). Vitamin D replenishment will be permitted, and participants may be re-screened once.

  - Hypercalcemia.

  - Elevated transaminases ≥ 3.0 x ULN.
  * Elevated TBL > 1.5 x ULN.
  * Albumin-adjusted serum calcium levels < 8.5 mg/dL or > 10.5 mg/dL.

Other Exclusions

* Female participants of childbearing potential unwilling to use protocol-specified method of contraception (see Appendix 5, Section 11.5) during treatment and for an additional 5 months after the last dose of Prolia®.
* Female participants who are breastfeeding or who plan to breastfeed while on study through 5 months after the last dose of Prolia®.
* Female participants planning to become pregnant while on study through 5 months after the last dose of Prolia®.
* Female participants of childbearing potential with a positive pregnancy test assessed at Screening by a serum pregnancy test.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant's and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Lumbar Spine BMD Percentage | At 12 months

SECONDARY OUTCOMES:
Change from Baseline in C-terminal Telopeptide (CTx) Expression | At 3, 6, 9, and 12 months
Change from Baseline in Procollagen Type 1 N-Telopeptide (P1NP) Expression | At 3, 6, 9, and 12 months
Change from Baseline in Hip and Femoral Neck BMD Percentage | At 6 and 12 months
Change from Baseline in Lumbar Spine BMD Percentage | At 6 months
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to 12 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a treatment, combination product, medical device, or procedure. TEAEs are any event that occurred after the participant received study treatment. Serious AEs (SAEs) are defined as any untoward medical occurrence that, meets at least 1 of the following serious criteria: immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- China (15):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou First Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Peoples Hospital, Shenzhen, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Huaian First Peoples Hospital, Huaian, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Pingxiang Peoples Hospital, Pingxiang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi An Jiaotong University, Xi'an, Shaanxi
  - Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Sichuan Provincial Peoples Hospital, Chengdu

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com